CLINICAL TRIAL: NCT05430061
Title: Impact of Slowly Digestible Carbohydrates on Gastric Emptying Rates
Brief Title: Crossover Trials Which Assessed Consumption of Slowly Digestible Carbohydrates for 21 Days on Gastric Emptying Rates
Acronym: INT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Principal Investigator / Distinguished professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1706019377
Record Dates: First submitted 2022-04-26; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: treatment (21 days of consumption of 30 g of raw corn starch) and control (21 days of consumption of maltodextrin)
Who Masked: Participant
Masking Description: Participants were not aware of the treatment recieved
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raw corn starch (Experimental): Raw corn starch is a slow digesting carbohydrate, corn starch, a commonly consumed food ingredient, considered GRAS (generally recognized as safe) CFR 182.70- 182.90 will be used as the test meal treatment. Participants will receive 21 individual containers of raw corn starch (30 g/container) and 21 cups of 4 oz unsweetened apple sauce. Participants will be asked to consume one starch container mixed in apple sauce at 10 a.m.; each day for 21 days.
  Interventions: Dietary Supplement: slowly digestible carbohydrate
- Maltodextrin DE-10 (Sham Comparator): Maltodextrin dextrose equivalent 10 is a fast digesting carbohydrate, is a non-sweet nutritive polymer that consists of D-glucose units linked primarily by [alpha]-1-4 bonds and that has a dextrose equivalent (D.E.) of less than 20. It is regarded as Generally Recognized as Safe (GRAS) by the U.S. Food and Drug Administration for direct use as a food ingredient (GRAS, 21CFR184.1444).DE-1 Maltodextrin is commercially available. Participants will receive 21 individual containers of maltodextrin (30 g/container) and 21 cups of 4 oz unsweetened apple sauce. Participants will be asked to consume one maltodextrin container mixed in apple sauce at 10 a.m.; each day for 21 days.
  Interventions: Dietary Supplement: slowly digestible carbohydrate

INTERVENTIONS:
Dietary Supplement: slowly digestible carbohydrate — carbohydrates with slow digestion rate have the capacity to induce slow gastric emptying time and potentially modify metabolic response and modulate postprandial glycemia.

SUMMARY:
To gain a better understanding about the conditioning effect of consumption of slowly digestible carbohydrate on gastric emptying rate, respiratory quotient and metabolic flexibility, this study will focus on monitoring change in gastric emptying with consumption of a single source of slowly digestible carbohydrate (30 g of raw corn starch) for 21 days and compared to a control (21 days of continious consumption of rapidly digesting carbohydrate maltodextrin).

DETAILED DESCRIPTION:
Corn starch, a commonly consumed food ingredient, considered GRAS (generally recognized as safe) CFR 182.70- 182.90 will be used as the test meal treatment fed to non-responding subjects (rapid gastric emptying rate after consumption of slowly digestible carbohydrate) for 1 month. Corn starch will be mixed with applesauce (200 g) and a small amount of xanthan gum (amount to be determined) (GRAS # 121) for palatability and viscosity, respectively.

In order to determine whether potential changes in gastric emptying time are induced by consumption of slowly digestible carbohydrates, a control group will be used. The control group will consume a meal composed applesauce (200 g) and xanthan gum with a fast digesting carbohydrate (30 g DE -1 maltodextrinpregelatinized starch). The product is commercially available and will be provided by Tate and Lyle under the brand name of Star-Dri 1. The general term "maltodextrin" is a non-sweet nutritive polymer that consists of D-glucose units linked primarily by [alpha]-1-4 bonds and that has a dextrose equivalent (D.E.) of less than 20. It is regarded as Generally Recognized as Safe (GRAS) by the U.S. Food and Drug Administration for direct use as a food ingredient (GRAS, 21CFR184.1444).DE-1 Maltodextrin is commercially available and will be provided by Tate and Lyle under the brand name of Star-Dri 1. Maltodextrin is a non-sweet nutritive saccharide polymer that consists of D-glucose units linked primarily by [alpha]-1-4 bonds and that has a dextrose equivalent (D.E.) of less than 20. It is regarded as Generally Recognized as Safe (GRAS) by the Food and Drug Administration for direct use as a food ingredient (GRAS, 21CFR184.1444). Ultimately, this study will help elucidate attributes of carbohydrate-based foods that can promote slow digestion and create a satiety feeling and promote weight management, which can then be implemented to develop foods with superior health benefits.

ELIGIBILITY:
Inclusion Criteria:

* normal body mass index (18.5 kg/m² < BMI < 25)
* healthy eating index score (<65)

Exclusion Criteria:

* gastrointestinal and cardiovascular disease
* food allergies or intolerances
* pregnancy
* smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Gastric half emptying time | 21 days of intervention
  Using a 13C octanoic acid breath test we assessed gastric emptying time using a non-invasive procedure

SECONDARY OUTCOMES:
Respiratory exchange ratio and metabolic flexibility | 21 days of intervention
  Using a portable, handheld device we assessed CO2 production after a consumption of a standardized meal. This device helped used determine RER and subsequent metabolic flexibility.
Height and Weight | Height and weight will only be entered at baseline.
  Height (in cm) and Weight (in Kg) will not be individually collected and will not be an outcome in the study. However, height and weight will be used by the algorithm using by the device (Lumen) to calculate RER. We do not expect to see changes in weight during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Hamaker, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing